CLINICAL TRIAL: NCT02071433
Title: Analgesic Efficacy of Saphenous Nerve Blockade for Outpatient Knee Anterior Cruciate Ligament Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, W ten Hoope, MD, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ACLS
Record Dates: First submitted 2014-02-24; First posted 2014-02-25 (Estimated); Last update posted 2017-01-26 (Estimated); Status verified 2017-01

CONDITIONS: Postoperative Analgesia for Anterior Cruciate Ligament Surgery of the Knee
Keywords: Saphenous nerve block; Adductor canal block; Anterior cruciate ligament; Pain management; Day care
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Saphenous nerve blockade (Experimental): Experimental treatment 15 mL of levobupivacaine 0.5%
  Interventions: Procedure: Saphenous nerve blockade
- Femoral nerve blockade (Active Comparator): Standard treatment 15 mL of levobupivacaine 0.5%
  Interventions: Procedure: Femoral nerve blockade

INTERVENTIONS:
Procedure: Saphenous nerve blockade
  Arms: Saphenous nerve blockade
Procedure: Femoral nerve blockade
  Arms: Femoral nerve blockade

SUMMARY:
The purpose of this study is to determine whether blockade of the saphenous nerve can provide the same degree of analgesia postoperatively for ACLS as a femoral nerve block without resulting motor blockade enhancing shortening of hospital stay en functional outcome.

ELIGIBILITY:
Inclusion Criteria:

* age 18-65 years
* ASA status I - III
* rupture of the anterior cruciate ligament.

Exclusion Criteria:

* contraindication for regional anesthesia
* allergy against local anesthetics
* BMI > 35
* pre-existing diagnosed neuropathy of the operated leg
* ingestion of strong opioids
* pregnancy or breastfeeding status
* History of significant cardiovascular disease (MI, CVA, peripheral vascular disease)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2014-03; Primary Completion 2017-07 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Readiness to discharge from day-care center in hours according to Post-Anesthetic Discharge Scoring System (PADSS).[ | 1 day

SECONDARY OUTCOMES:
Motor block | 2 days
Pain (VAS) | 2 days
Sensory blockade extent | 1 Day
Time to rescue analgesic and post operative opioid consumption | 1 Day
Overall Benefit of Analgesia Score (OBAS) | 6 weeks
SF-12 score | 12 weeks
KOOS-score | 12 weeks
IKDC-score | 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Academic Medical Centre Amsterdam, Amsterdam, Netherlands